CLINICAL TRIAL: NCT00344032
Title: Phase IIIb, Double-blind, Randomized, Controlled Study to Evaluate the Immunogenicity and Safety of GSK Biologicals' HPV-16/18 VLP/AS04 Vaccine Administered Intramuscularly at 0, 1, 6 Months in Healthy Indian Female Subjects Aged 18-35 Yrs
Brief Title: Evaluation of the Immune and Safety Response of GlaxoSmithKline (GSK) Biologicals' HPV Vaccine in Healthy Indian Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 104479
Record Dates: First submitted 2006-06-23; First posted 2006-06-26 (Estimated); Results first posted 2009-12-15 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2016-11

CONDITIONS: Infections, Papillomavirus
Keywords: Double-blind; Human Papillomavirus; Phase IIIb; Controlled; Randomized; India
MeSH Terms: conditions — Papillomavirus Infections | interventions — human papillomavirus vaccine, L1 type 16, 18

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Cervarix (Experimental): Subjects who received 3 doses of HPV-16/18 VLP/AS04 Vaccine (Cervarix TM) (at 0, 1, 6 months).
  Interventions: Biological: HPV-16/18 VLP/AS04 Vaccine (Cervarix TM)
- Placebo (Placebo Comparator): Subjects who received 3 doses of Placebo (at 0, 1, 6 months).
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Arms: Placebo
Biological: HPV-16/18 VLP/AS04 Vaccine (Cervarix TM) — Three doses of vaccine administered intramuscularly according to a 0, 1, 6-month schedule.
  Other Names: GSK Biologicals' HPV-16/18 VLP/AS04 vaccine
  Arms: Cervarix

SUMMARY:
Human papillomavirus infection has clearly been recognized as the cause of cervical cancer. Indeed, the infection of the cervix by certain oncogenic types of HPV, if not cleared , can lead over time to cervical cancer in women . This study will evaluate the immune response induced by the HPV-16/18 L1/AS04 vaccine and the safety of the vaccine.

The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

All subjects must satisfy the following criteria at study entry:

* Subjects who the investigator believes that they can and will comply with the requirements of the protocol should be enrolled in the study.
* A female between, and including, 18 and 35 years of age at the time of the first vaccination.
* Written informed consent obtained from the subject.
* Healthy subjects as established by medical history and clinical examination before entering into the study.
* Subjects must have a negative urine pregnancy test.
* Subjects of childbearing potential at the time of study entry must be abstinent or must be using adequate contraceptive precautions for 30 days prior to vaccination and must agree to continue such precautions for two months after completion of the vaccination series.

Exclusion Criteria:

The following criteria should be checked at the time of study entry. If any apply, the subject must not be included in the study:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine/ control within 30 days preceding the first dose of study vaccine/ control, or planned use during the study period.
* Pregnant or breastfeeding.
* Planning to become pregnant or likely to become pregnant.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose.
* Planned administration/administration of a vaccine not foreseen by the study protocol within 30 days (Days 1 to 30) before and 30 days (Day 0- Day 29) after the first dose of vaccine. Administration of routine meningococcal, hepatitis B, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus-containing vaccine up to 8 days before the first dose of study vaccine is allowed.
* Previous administration of components of the investigational vaccine.
* Previous vaccination against HPV.
* Any medically diagnosed or suspected immunodeficient condition based on medical history and physical examination.
* History of allergic disease, suspected allergy or reactions likely to be exacerbated by any component of the study vaccines.
* Hypersensitivity to latex.
* Known acute or chronic, clinically significant neurologic, hepatic or renal functional pulmonary, cardiovascular abnormality, as determined by previous physical examination or laboratory tests.
* History of chronic condition(s) requiring treatment.
* Administration of immunoglobulins and/or any blood product within three months preceding the first dose of study vaccine/ control or planned administration during the study period. Enrolment will be deferred until condition is resolved.
* Acute disease at the time of enrolment. Acute disease is defined as the presence of a moderate or severe illness with or without fever.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 354 (Actual)
Dates: Start 2006-07-28; Primary Completion 2007-12-01 (Actual); Study Completion 2007-12-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (4):
- India (4):
  - GSK Investigational Site, Chandigarh
  - GSK Investigational Site, Kolkata
  - GSK Investigational Site, Mumbai
  - GSK Investigational Site, New Delhi

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Bhatla N, Suri V, Basu P, Shastri S, Datta SK, Bi D, Descamps DJ, Bock HL; Indian HPV Vaccine Study Group. Immunogenicity and safety of human papillomavirus-16/18 AS04-adjuvanted cervical cancer vaccine in healthy Indian women. J Obstet Gynaecol Res. 2010 Feb;36(1):123-32. doi: 10.1111/j.1447-0756.2009.01167.x. PMID 20178538
- [Background] Verstraeten T, Descamps D, David MP, Zahaf T, Hardt K, Izurieta P, Dubin G, Breuer T. Analysis of adverse events of potential autoimmune aetiology in a large integrated safety database of AS04 adjuvanted vaccines. Vaccine. 2008 Dec 2;26(51):6630-8. doi: 10.1016/j.vaccine.2008.09.049. PMID 18845199
- [Derived] Bergman H, Henschke N, Arevalo-Rodriguez I, Buckley BS, Crosbie EJ, Davies JC, Dwan K, Golder SP, Loke YK, Probyn K, Petkovic J, Villanueva G, Morrison J. Human papillomavirus (HPV) vaccination for the prevention of cervical cancer and other HPV-related diseases: a network meta-analysis. Cochrane Database Syst Rev. 2025 Nov 24;11(11):CD015364. doi: 10.1002/14651858.CD015364.pub2. PMID 41276263
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Informed Consent Form: 104479 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 104479 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 104479 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 104479 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 104479 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 104479 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cervarix | Placebo
Started | 176 | 178
Completed | 162 | 168
Not Completed | 14 | 10
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 6 | 2
Not completed — Lost to Follow-up | 4 | 6
Not completed — Physician Decision | 4 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cervarix | Placebo | Total
Number analyzed (Participants) | 176 | 178 | 354
Age, Continuous [Mean (Standard Deviation); unit: Years] | 28.5 (4.70) | 28.5 (4.97) | 28.5 (4.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 176 | 178 | 354
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Who Seroconverted for Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Seroconversion is defined as the appearance of antibodies with titers greater than or equal to the predefined cut-off value in the serum of subjects seronegative before vaccination. Cut-off values assessed include 8 enzyme-linked immunosorbent assay units per milliliter (EL.U/mL) for anti-HPV-16 antibodies and 7 EL.U/mL for anti-HPV-18 antibodies.
Time Frame: At Month 7
Population: Analysis was performed on initially seronegative subjects from the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix | Placebo
Number analyzed (Participants) | 124 | 139
Participants
  Anti-HPV-16 | 124 | 16
  Anti-HPV-18: number analyzed (Participants) | 117 | 124
  Anti-HPV-18 | 117 | 4

2. Secondary Outcome: Titers of Anti-human Papilloma Virus 16 (Anti-HPV-16) and Anti-human Papilloma Virus 18 (Anti-HPV-18) Antibodies
Description: Titers are given as Geometric Mean Titers (GMTs) expressed as Enzyme-linked Immunosorbent Assay Units Per Milliliter (EL.U/mL).
Time Frame: At Months 0 and 7
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for analysis of immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: EL.U/mL
Arm/Group | Cervarix | Placebo
Number analyzed (Participants) | 148 | 158
EL.U/mL
  Anti-HPV-16 (Month 0) | 5.4 [4.7 to 6.1] | 4.9 [4.4 to 5.5]
  Anti-HPV-16 (Month 7): number analyzed (Participants) | 148 | 156
  Anti-HPV-16 (Month 7) | 9813.8 [8605.4 to 11191.9] | 6.0 [5.1 to 7.0]
  Anti-HPV-18 (Month 0): number analyzed (Participants) | 148 | 156
  Anti-HPV-18 (Month 0) | 4.7 [4.2 to 5.2] | 4.6 [4.2 to 5.1]
  Anti-HPV-18 (Month 7): number analyzed (Participants) | 148 | 154
  Anti-HPV-18 (Month 7) | 4030.1 [3544.0 to 4582.8] | 4.9 [4.3 to 5.5]

3. Secondary Outcome: Number of Subjects Reporting Solicited Symptoms
Description: Solicited local symptoms assessed include pain, redness and swelling. Solicited general symptoms assessed include arthralgia, fatigue, fever, gastro-intestinal symptoms, headache, myalgia, rash and urticaria.
Time Frame: During the 7 days (Days 0 - 6) after each vaccination
Population: Analysis was performed on the Total Vaccinated Cohort, on subjects with available data.
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix | Placebo
Number analyzed (Participants) | 171 | 174
Participants
  Pain | 137 | 105
  Redness | 56 | 24
  Swelling | 69 | 35
  Arthralgia | 19 | 16
  Fatigue | 84 | 83
  Fever (above 37.5 degree Celsius) | 51 | 48
  Gastro-intestinal symptoms | 25 | 28
  Headache | 72 | 71
  Myalgia | 10 | 11
  Rash | 5 | 8
  Urticaria | 4 | 6

4. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events (AEs)
Description: Unsolicited adverse event = Any adverse event (AE) reported in addition to those solicited during the clinical study. Also any "solicited" symptom with onset outside the specified period of follow-up for solicited symptoms was reported as an unsolicited adverse event.
Time Frame: Within 30 days (Days 0 - 29) after each vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix | Placebo
Number analyzed (Participants) | 176 | 178
Participants | 20 | 26

5. Secondary Outcome: Number of Subjects Reporting Unsolicited Adverse Events as New Onset Chronic Diseases (NOCDs) and Other Medically Significant Adverse Events (AEs)
Description: NOCDs assessed include e.g. autoimmune disorders, asthma, type I diabetes. Medically significant AEs assessed include AEs prompting emergency room or physician visits that are not related to common diseases or SAEs that are not related to common diseases.
Time Frame: Throughout the study period (up to Month 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix | Placebo
Number analyzed (Participants) | 176 | 178
Participants
  NOCDs | 0 | 2
  Medically Significant AEs | 13 | 24

6. Secondary Outcome: Number of Subjects Reporting Serious Adverse Events
Description: Serious adverse events assessed include medical occurrences that results in death, is life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Throughout the study period (up to Month 7)
Measure: Count of Participants; unit: Participants
Arm/Group | Cervarix | Placebo
Number analyzed (Participants) | 176 | 178
Participants | 2 | 4

ADVERSE EVENTS:
Description: Events collected by systematic assessment are reported for subjects with a symptom diary card available.
  Events collected by non-systematic method are reported for the Total Vaccinated Cohort
Arm/Group | Cervarix | Placebo
Serious Adverse Events (participants affected / at risk) | 2/176 | 4/178
Other Adverse Events (participants affected / at risk) | 153/176 | 132/178
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix (N=176) | Placebo (N=178)
Aborption spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bronchogenic cyst (Congenital, familial and genetic disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Lymph node tuberculosis (Infections and infestations) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cervarix (N=176) | Placebo (N=178)
Pain (General disorders) | 137 | 105
Redness (General disorders) | 56 | 24
Swelling (General disorders) | 69 | 35
Arthralgia (General disorders) | 19 | 16
Fatigue (General disorders) | 84 | 83
Fever (above 37.5 degree Celsius) (General disorders) | 51 | 48
Gastro-intestinal symptoms (General disorders) | 25 | 28
Headache (General disorders) | 72 | 71
Myalgia (General disorders) | 10 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.